CLINICAL TRIAL: NCT04978285
Title: Association of Postoperative Anaemia With Patient-centred Outcomes
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: 544/12
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2021-07

CONDITIONS: Anemia After Surgery
Keywords: anemia; complications; hemoglobin; iron; patient-centered outcome; surgery
MeSH Terms: conditions — Anemia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative anemia: All patients enrolled in the RELIEF trial in which a postoperative Day 1-3 hemoglobin concentration was measured. Anaemia will be defined according to the World Health Organisation definition (males Hb <130 g/L, and female Hb <120 g/L).
  Interventions: Other: Anemia
- No postoperative anemia: All patients enrolled in the RELIEF trial in which a postoperative Day 1-3 hemoglobin concentration was measured. No anaemia will be defined according to the World Health Organisation definition (males Hb ≥130 g/L, and females Hb ≥120 g/L).
  Interventions: Other: Anemia

INTERVENTIONS:
Other: Anemia — Depends on Day 3 Hb result
  Other Names: Observational

SUMMARY:
Primary aim - To investigate the relationship between postoperative anaemia and patient-centred outcomes after major abdominal surgery.

Secondary aim - To determine whether a more liberal perioperative IV fluid strategy increases the risk of postoperative anaemia (haemodilution).

Hypothesis: Adults with anaemia in the immediate postoperative period following major abdominal surgery have a poorer quality of recovery and higher risk of complications, leading to poor disability-free survival when compared with patients without postoperative anaemia.

DETAILED DESCRIPTION:
The consequences of postoperative anemia remain unclear. Postoperative anaemia is more likely if there is pre-existing anemia, but also increased perioperative blood loss, frequent blood sampling, excess IV fluids (leading to hemodilution), sepsis, and inadequate nutritional intake after surgery. A nadir in Hb concentration is most often observed within the first 3-4 days after surgery. Postoperative anemia is believed to have deleterious effects on patient outcomes, including prolonged hospital stay, increased postoperative complications, and perhaps poor survival, but there is very little data to support this belief.

A recent consensus statement suggested that all patients recovering from major surgery (defined as blood loss > 500 ml or lasting > 2 h) and either had preoperative anemia or moderate-to-severe blood loss during surgery must be screened for anemia after surgery. Furthermore, this consensus group recommended that patients recovering from uncomplicated major surgery should have their Hb concentration measured for at least 3 days after surgery to detect anemia. As outlined above, this is problematic if there is fluid retention.

The role of IV iron for the treatment of postoperative anemia is unclear, with the most recent systematic review concluding that neither oral nor IV iron had a significant effect on patient quality of life or functional outcomes following surgery. A diagnosis of iron deficiency is very difficult in the postoperative period because the acute phase inflammatory response results in spuriously elevated ferritin levels, and several studies have demonstrated oral iron therapy is ineffective in this setting.

The investigators propose a study to investigate the incidence, extent, and outcomes of patients with anemia after major surgery, including an assessment of the amount of IV fluids administered in the immediate perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) undergoing elective major surgery and providing informed consent
2. All types of open or lap-assisted abdominal or pelvic surgery with an expected duration of at least 2 hours, and an expected hospital stay of at least 3 days
3. At increased risk of postoperative complications, as defined by any of the following criteria:

   1. age ≥70 years
   2. known or documented history of coronary artery disease
   3. known or documented history of heart failure
   4. diabetes currently treated with an oral hypoglycemic agent and/or insulin
   5. preoperative serum creatinine >200 micromol/L (>2.8 mg/dl)
   6. morbid obesity (BMI ≥35 kg/m2)
   7. preoperative serum albumin <30 g/L
   8. anaerobic threshold (if done) <12 mL/kg/min
   9. or two or more of the following risk factors:

      * ASA 3 or 4
      * chronic respiratory disease
      * obesity (BMI 30-35 kg/m2)
      * aortic or peripheral vascular disease
      * preoperative Hb <100 g/L
      * preoperative serum creatinine 150-199 micromol/L (>1.7 mg/dl)
      * anerobic threshold (if done) 12-14 mL/kg/min

Exclusion Criteria:

1. Urgent or time-critical surgery
2. ASA physical status 5 - such patients are not expected to survive with or without surgery, and their underlying illness is expected to have an overwhelming effect on outcome (irrespective of fluid therapy)
3. Chronic renal failure requiring dialysis
4. Pulmonary or cardiac surgery - different pathophysiology, and thoracic surgery typically have strict fluid restrictions
5. Liver resection - most units have strict fluid/CVP limits in place and won't allow randomisation
6. Minor or intermediate surgery, such as laparoscopic cholecystectomy, transurethral resection of the prostate, inguinal hernia repair, splenectomy, closure of colostomy - each of these are typically "minor" surgery with minimal IV fluid requirements, generally low rates of complications and mostly very good survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, elective major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Persistent disability or death by 90 days | 90 days after surgery
  Defined as a World Health Organization Disability Assessment Schedule 2.0 (WHODAS) score of at least 24 points (on the 48-point scale) at both 30 and 90 days postoperatively, reflecting a disability level of at least 25% and being the threshold point between "disabled" and "not disabled" as per WHO guidelines. Disability was assessed by the participant, but if unable then we used the proxy's report.

SECONDARY OUTCOMES:
Death: all-cause mortality at 90 days, then up to 12 months after surgery | 1 year
A composite (pooled) and individual septic complications: sepsis, surgical site infection, anastomotic leak, and pneumonia | 30 days
Sepsis: using Centers for Disease Control and Prevention (CDC) with National Healthcare Safety Network (NHSN) criteria | 30 days
Surgical site infection | 30 days
  CDC criteria
Pneumonia | 30 days
  The presence of new and/or progressive pulmonary infiltrates on chest radiograph plus two or more of the following:
  i. Fever ≥ 38.5°C or postoperative hypothermia <36°C ii. Leucocytosis ≥ 12,000 WBC/mm3 or leucopenia < 4,000 WBC/mm3 iii. Purulent sputum and/or iv. New onset or worsening cough or dyspnea.
Anastomotic leak | 30 days
  A defect of the intestinal wall at the anastomotic site (including suture and staple lines of neorectal reservoirs) leading to a communication between the intra- an extra luminal compartments.
Acute kidney injury | 30 days
  According to The Kidney Disease: Improving Global Outcomes (KDIGO) group criteria, but not urine output - for Stage 2 or worse AKI defined as at least 2-fold increase in creatinine, or estimated GFR decrease >50%
Unplanned admission to ICU within 30 days of surgery | 30 days
ICU stay | 30 days
  Total days - additive, including initial ICU admission and readmission times up to Day 30
Hospital stay | 30 days
  Total -additive, from the start (date, time) of surgery until actual hospital discharge , plus readmission(s) up to Day 30
Quality of recovery | Postoperative Days 3 and 30
  QoR-15 scale score
Hospital re-admission | At 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Consider, on request

REFERENCES:
- [Background] Myles PS, Bellomo R, Corcoran T, Forbes A, Peyton P, Story D, Christophi C, Leslie K, McGuinness S, Parke R, Serpell J, Chan MTV, Painter T, McCluskey S, Minto G, Wallace S; Australian and New Zealand College of Anaesthetists Clinical Trials Network and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus Liberal Fluid Therapy for Major Abdominal Surgery. N Engl J Med. 2018 Jun 14;378(24):2263-2274. doi: 10.1056/NEJMoa1801601. Epub 2018 May 9. PMID 29742967
- [Derived] Myles PS, Richards T, Klein A, Wood EM, Wallace S, Shulman MA, Martin C, Bellomo R, Corcoran TB, Peyton PJ, Story DA, Leslie K, Forbes A; RELIEF Trial Investigators. Postoperative anaemia and patient-centred outcomes after major abdominal surgery: a retrospective cohort study. Br J Anaesth. 2022 Sep;129(3):346-354. doi: 10.1016/j.bja.2022.06.014. Epub 2022 Jul 15. PMID 35843746

DOCUMENTS (2):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT04978285/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT04978285/SAP_001.pdf